CLINICAL TRIAL: NCT06308159
Title: An Open-label Clinical Trial of Ex Vivo Beta-globin Lentiviral Vector Transduction of Autologous CD34+HSPCs (Vebeglogene Autotemcel) for the Treatment of Transfusion Dependent Beta-thalassemia Patients
Brief Title: An Open-label Study of a Gene Therapy Product (Vebeglogene Autotemcel) in Transfusion Dependent Beta-Thalassemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lantu Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT02-101
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vebeglogene autotemcel (Experimental): One-time infusion of≥5×10^6/kg beta-globin lentiviral vector transduced HSPCs
  Interventions: Drug: Vebeglogene autotemcel

INTERVENTIONS:
Drug: Vebeglogene autotemcel — Autologous HSPCs transduced with self-inactivating lentiviral vector encoding functional HBB gene and resuspended in cryopreservative solution in the final immediate container for the intended medical use.
  Other Names: Beta-globin lentiviral vector transduced autologous HSPCs

SUMMARY:
This is an interventional study to evaluate the safety and efficacy of autologous Hematopoietic Stem and Progenitor Cells (HSPCs) transduced with lentiviral vector encoding functional hemoglobin subunit beta (HBB) gene in patients with transfusion-dependent beta-thalassemia.

DETAILED DESCRIPTION:
The participant's autologous HSPCs will be transduced with the self-inactivating lentiviral vector, carrying the functional HBB gene.

Study duration per participant is approximately 27 months including an approximately 30-day screening/baseline period, an approximately 60-day mobilization and product manufacture, an approximately 10-day myeloablative conditioning, 1 treatment day, and an approximately 24-month study observation period.

The endpoints will be used to assess the safety and efficacy profiles in patients with transfusion-dependent beta-thalassemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients or parent(s)/legal guardian(s) willing and able to complete the informed consent process and comply with study procedures and visit schedules.
* Diagnosis of beta-thalassemia and a history of RBCs transfusions.
* Documented baseline, or pretransfusion, Hb≤7 g/dL.
* Availability of an adequate and well-documented transfusion history.

Exclusion Criteria:

* Active bacterial, viral, fungal, or parasitic infection.
* A white blood cell (WBC) counts<3×10^9/L, and/or platelet counts<100×10^9/L not related to hypersplenism.
* Uncorrected bleeding disorder.
* Presence of severe diseases that judged not compatible with the study procedures, such as severe hepatic disease, kidney disease, lung disease, and/or cardiovascular disease.
* Uncontrolled seizure disorder.
* Any evidence of severe iron overload that, in the investigator's opinion, warrants exclusion.
* Prior autologous hematopoietic stem cell transplantation.
* Prior receipt of gene therapy.

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-05-11 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Time and duration of the subject's hemoglobin (Hb)≥9.0 g/dL without receiving red blood cell infusion | From baseline to Month 24

SECONDARY OUTCOMES:
The prevalence and severity of adverse events (AEs) and serious adverse events (SAEs) | From baseline to Month 24
  Participants are monitored for safety from baseline up to the end of the follow-up period.
The reduction of red blood cells (RBCs) transfusion requirement after product infusion compared to previous transfusion records | From infusion to Month 24
  The annual number of RBCs transfusions prior to product infusion will be compared to the annual number of RBCs transfusions post-infusion, and the requirement reduction duration should be reported.
Number of days required to achieve successful neutrophil and platelet engraftment | From infusion to Month 24
  Neutrophil engraftment is defined as the time to the first of 3 consecutive days of absolute neutrophil counts (ANC)≥0.5×10^9/L post-infusion without transfusion. Platelet engraftment is defined as the time to the first of 3 consecutive days of platelet values≥20×10^9/L post-infusion without transfusion.
Vector copy number (VCN) in peripheral blood over time | From baseline to Month 24
  Quantification of the lentiviral vector copy number in individual peripheral blood cells will be conducted to measure the transduction of HSPCs.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan
  - Kunming Hope of Health Hospital, Kunming, Yunnan